CLINICAL TRIAL: NCT00992316
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Parallel Group, Dose Escalation Study To Investigate The Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-04531083 In Healthy Male Subjects
Brief Title: To Investigate The Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-04531083 In Healthy Male Subjects
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: B1351001
Record Dates: First submitted 2009-09-04; First posted 2009-10-09 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Pain
Keywords: Inflammatory pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pf-04531083: To Investigate The Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-04531083 In Healthy Male Subjects
  Interventions: Drug: PF-04531083

INTERVENTIONS:
Drug: PF-04531083 — solution. doses to be selected based upon safety/tolerability/PK at preceeding dose

SUMMARY:
The purpose of the study is to investigate the safety, toleration and pharmacokinetics of single oral doses of PF-04531083 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* young
* healthy
* male

Exclusion Criteria:

* elderly
* unhealthy
* female

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young, healthy male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and toleration: adverse events, supine and standing vital sign measurements,telemetry, 12-lead ECGs, blood and urine safety tests | up to 48 hours
Plasma: Cmax, Tmax, AUClast, AUCinf, AUC0-24, CL/F and t½ for PF-04531083 | 240 hours post dose
Cmax, Tmax, AUClast, AUCinf and t½ for PF-04335882 | 240 hours post dose
Urine: Aet (amount excreted in urine), Aet% and CLr (for selected doses dependent on the emerging pharmacokinetic profile of PF-04531083, PF-04335882 and O-desmethyl metabolite (PF-04959926))where t = 48 hours. | 240 hours post dose

SECONDARY OUTCOMES:
No secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351001&StudyName=To%20Investigate%20The%20Safety%2C%20Toleration%20And%20Pharmacokinetics%20Of%20Single%20Oral%20Doses%20Of%20PF-04531083%20In%20Healthy%20Male%20Subjects